CLINICAL TRIAL: NCT03185780
Title: Impact of Complementary/Integrative Medicine Treatments on Patients With Brain Cancer: A Pilot Study
Brief Title: Complementary/Integrative Medicine for Brain Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to attain funding
Sponsor: The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, Noah Samuels, Medical Director, Tal Center for Integrative Oncology, Institute of Oncology, The Chaim Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ChaimShebaMC
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Quality of Life; Chemotherapeutic Toxicity; Radiation Toxicity
Keywords: complementary/integrative medicine; glioblastoma; quality of life; adherence
MeSH Terms: conditions — Radiation Injuries; Glioblastoma | interventions — Acupuncture Therapy; Acupressure

STUDY DESIGN:
Intervention Model Description: Patients with high grade glioma undergoing adjuvant (post-surgical) chemo-radiation treatment will be treated with acupuncture and/or touch therapies, this in parallel to their conventional treatment regimen. The primary study outcome will be the scores on four Patient-Reported Outcome Measures (PROMs): the Measure Yourself Concerns and Wellbeing (MYCAW) study tool; the Functional Assessment of Cancer Therapy, Brain Cancer (FACT-Br) questionnaire; the Edmonton Symptom Assessment Scale (ESAS); and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-c30). Secondary study outcomes will include the safety of the complementary medicine treatments, and adherence to the planned oncology treatment regimen, as measured by the Relative Dose Intensity (RDI) calculation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients will be treated with acupuncture and/or touch therapies, this in parallel to their chemo-radiation regimen. These treatments will be administered twice-weekly during active chemo-radiation treatment (6 weeks), followed by once-weekly treatment throughout the remainder of the study period (6 months)
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture: the insertion of use of ultra-fine needles (diameter 0.18 - 0.30mm) into designated "acupoints" in the skin, along the limbs and trunk areas.
  Reflexology: The massage + application of localized pressure on designated points along the plantar aspect of the feet.
  Shiatsu: The application of localized pressure along designated points (similar to "acupoints") along the limbs and trunk areas.
  Other Names: Touch Therapy - reflexology or Shiatsu

SUMMARY:
Nearly a quarter of a million patients are diagnosed each year with tumors of the central nervous system, a third of them malignant. The most common malignant tumor of the brain is the high grade glioma( HGG), whose treatment begins with surgical resection of the tumor, followed by a combined chemo-radiation regimen, with the drug Temodal (temozolomide). This treatment is often accompanied by toxic effects (e.g., nausea, headache, constipation, weakness/fatigue, and others), with treatment of these effects limited in their effectiveness and safety. Complementary medicine treatments such as acupuncture and touch therapies (reflexology, Shiatsu, etc.) have been researched and found to be both safe and effective for some of the toxic effects of oncology treatment regimens.

The present pilot study is set to examine the impact of complementary medicine on the toxic effects of the conventional treatment for HGG. The study will include 40 patients and will last for two years, during which patients will be treated with acupuncture and/or touch therapies, this in parallel to their chemo-radiation regimen. The primary study outcome will be the scores on four Patient-Reported Outcome Measures (PROMs): the Measure Yourself Concerns and Wellbeing (MYCAW) study tool; the Functional Assessment of Cancer Therapy, Brain Cancer (FACT-Br) questionnaire; the Edmonton Symptom Assessment Scale (ESAS); and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-c30). Secondary study outcomes will include the safety of the complementary medicine treatments, and adherence to the planned oncology treatment regimen, as measured by the Relative Dose Intensity (RDI) calculation.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 18 years and older
* diagnosed with high grade glioma (stage III-IV)
* following surgical intervention (tumor resection)
* prior to chemo-radiation treatment
* signing of informed consent form

Exclusion Criteria:

* inability/unwillingness to sign informed consent form
* unwillingness of treating oncologist to allow participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure Yourself Concerns and Wellbeing (MYCAW) study tool | 6 months
  Patient-Reported Outcome Measure - Quality of Life Assessment
Functional Assessment of Cancer Therapy, Brain Cancer (FACT-Br) questionnaire | 6 months
  Patient-Reported Outcome Measure - Quality of Life Assessment
Edmonton Symptom Assessment Scale (ESAS) | 6 months
  Patient-Reported Outcome Measure - Quality of Life Assessment
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-c30) | 6 months
  Patient-Reported Outcome Measure - Quality of Life Assessment

SECONDARY OUTCOMES:
Adverse effects attributed to the complementary/integrative medicine treatments | 6 months
  Relates to the safety of the complementary medicine treatments
RDI - relative dose intensity | 6 months
  Reflects adherence to the conventional chemo-radiation treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Noah Samuels, MD, Principal Investigator — Tal Center for Integrative Oncology, Institute of Oncology, Chaim Sheba Medical Center, Israel

IPD SHARING:
Plan to Share IPD: Undecided